# **Cover Page for Protocol**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT04007107 |
| Sponsor trial ID: | INS-4582 |
| Official title of study: | A TRIAL TO COMPARE THE INJECTION SITE PAIN EXPERIENCE OF 0.25 MG SEMAGLUTIDE SC ADMINISTERED BY 2 DIFFERENT PRODUCTS |
| Document date: | 17 March 2020 |

| Clinical Trial Report Appendix 16.1.1 Status: Final Page: 1 of 59 | 1 | 1 | CONFIDENTIAL | 1.0<br>Final | Novo Nordisk |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

# 16.1.1 Protocol

# **List of contents**

| CLINICAL STUDY PROTOCOL, INS-4582/ | , VERSION 2.0, 21 JUN 2019 2 |
|------------------------------------|------------------------------|
| 16.1.1.1 Filenote 03-Jun-2019 | |

Redacted protocol Includes redaction of personal identifiable information only.

#### **CLINICAL STUDY PROTOCOL**

# A TRIAL TO COMPARE THE INJECTION SITE <u>PAIN</u> EXPERIENCE OF 0.25 MG SEMAGLUTIDE SC ADMINISTERED BY 2 DIFFERENT PRODUCTS

CONFIDENTIAL

Sponsor code: INS-4582

code:

EudraCT number: 2019-002284-10 Universal Trial Number: U1111-1233-9590

Comparison of injection site *pain* experience for semaglutide sc

Investigational product: Semaglutide
Clinical phase: Phase 3b 2 study
Indication to be studied: Not applicable

Sponsor: Novo Nordisk A/S

Novo Allé

DK-2880 Bagsvaerd

Denmark

Contract Research Organization and Clinical Site:

Principal Investigator:

Phone: Fax: E-mail:

<u>Version 2.0, 21 Jun 2019</u> Version 1.0, 03 Jun 2019

This study will be performed in compliance with the principles of Good Clinical Practice.

# SPONSOR AUTHORIZATION OF CLINICAL STUDY PROTOCOL

The Sponsor and the Contract Research Organization agree to conduct the study as outlined in this clinical study protocol. Any modification of the clinical study protocol must be agreed upon by the Sponsor and the Contract Research Organization and must be documented in writing.

| Name/Position: | Date: | Signature: |
|------------------------------------|-------|------------|
| Sponsor: Novo Nordisk A/S | | |
| Senior International Trial Manager | | |
| International Project Statistician | | |
| Medical Specialist | | |

# AUTHORIZATION OF CLINICAL STUDY PROTOCOL BY CONTRACT RESEARCH ORGANIZATION

The Sponsor and the Contract Research Organization agree to conduct the study as outlined in this clinical study protocol. Any modification of the clinical study protocol must be agreed upon by the Sponsor and the Contract Research Organization and must be documented in writing.

| Name/Position: | <u>Date:</u> | <u>Signature:</u> |
|---------------------------------|--------------|-------------------|
| Contract Research Organization: | | |

### **CONTACT INFORMATION**

# **Sponsor**

Novo Nordisk A/S Novo Allé DK-2880 Bagsvaerd Denmark

# Sponsor's Contact

| Trial Operations, Insulin & Devices |
|--------------------------------------------------|
| Phone: |
| E-mail: |
| Sponsor's Medical Specialist |
| Medical & Science, Devices & Titration |
| Phone: |
| email: |
| Contract Research Organization and Clinical Site |
| Phone: |
| Fax: |
| Clinical Site Contacts |
| Phone: |
| Fax: |
| E-mail: |
| Phone: |
| Fax: |
| E-mail: |

# Clinical Laboratory Phone: Fax: Medical Screening Centers





Phone:

# **SUMMARY OF CHANGES**

<u>The following changes have been introduced in this Version 2.0 of the protocol and are given as a combination of double underlined and italic text. Deleted text is given as double strikethrough.</u>

- <u>In the study title and other sections of the protocol, the word 'pain' has been added between the words 'injection site' and 'experience' for clarification.</u>
- The clinical phase of the study has been changed from Phase 3b to Phase 2.
- <u>The language on subject numbering has been changed.</u>

#### The changes can be found in:

- <u>Title Page</u>
- Synopsis
- Section 1.3, Study Rationale
- Section 2, OBJECTIVES
- Section 4.1.1, Type of Study
- <u>Section 4.4.3, Method of Assigning Subjects to Treatment Groups</u>

#### **SYNOPSIS**

#### **Study Title**

A TRIAL TO COMPARE THE INJECTION SITE  $\underline{PAIN}$  EXPERIENCE OF 0.25 MG SEMAGLUTIDE SC ADMINISTERED BY 2 DIFFERENT PRODUCTS

#### **Short Study Title**

Comparison of injection site *pain* experience for semaglutide sc

**Study Codes** 

Sponsor code : INS-4582

code :

EudraCT number : 2019-002284-10 Universal Trial Number : U1111-1233-9590

**Sponsor** 

Novo Nordisk A/S, Novo Allé, DK-2880 Bagsvaerd, Denmark

Sponsor's contact :

#### **Contract Research Organization and Clinical Site**

#### **Principal Investigator**

<u>Clinical Phase</u> <u>: 2</u>

#### **Objectives**

The primary objective is to compare, in healthy subjects, the injection site <u>pain</u> experience of a single dose of 0.25 mg semaglutide subcutaneously (sc), given as the DV3396 product, to that of the PDS290 product.

#### **Endpoints**

Primary Endpoint

| Endpoint Title | Time Frame | Unit |
|---|---|---|
| Intensity of injection site pain | 1 min after each injection (Day 1) | mm on a 100-mm horizontal |
| | | visual-analogue scale (where |
| | | 0 mm= no pain, 100 mm = |
| | | unbearable pain) |

#### **Exploratory Endpoints**

| Endpoint Title | Time Frame | Unit |
|---|---|---|
| Categorical assessment of | Immediately after rating of | 6-point scale (none – very mild – |
| injection site pain | intensity of injection site pain, ie, | mild – moderate – severe – very |
| | after 1 min plus the time it takes | severe) |
| | to complete the rating of intensity | |
| | of injection site pain by visual | |
| | analogue scale (Day 1) | |
| Moderate or more injection site | Dichotomous variable based on | Yes = moderate, severe, very |
| pain | categorical assessment of | severe |

| Endpoint Title | Time Frame | Unit |
|---|---|---|
| - | intensity of injection site pain | No = none, very mild, mild |
| | (Day 1) (item above) | |
| Quality of pain | Immediately after categorical | Pain quality items on modified |
| | assessment of intensity of | SF-MPQ-2 inventory (select all |
| | injection site pain, ie, after 1 min | that apply): |
| | plus the time it takes to complete | Throbbing pain □ |
| | the rating of intensity of injection | Shooting pain □ |
| | site pain and the categorical rating of intensity of injection site | Stabbing pain □ |
| | pain (Day 1) | Sharp pain □ |
| | pair (Bay 1) | Cramping pain □ |
| | | Gnawing pain □ |
| | | Hot-burning pain □ |
| | | Aching pain □ |
| | | Heavy pain □ |
| | | Tender □ |
| | | Splitting pain □ |
| | | Tiring-exhausting □ |
| | | Sickening |
| | | Fearful Description and Formula Frequency Freq |
| | | Punishing-cruel □ |
| | | Electric-shock pain □ |
| | | Cold-freezing pain □ |
| | | Piercing |
| Duration of pain | From time of injection until | min and sec |
| Comparative pain experience | cessation of pain (Day 1) After pain has ended after the | 5-point scale (the last injection |
| Comparative pain expensive | last injection (Day 1) | hurt much more than the first |
| | last injection (Day 1) | injection – the last injection hurt |
| | | more than the first injection – |
| | | they hurt about the same |
| | | [includes: none of the injections |
| | | hurt] – the last injection hurt less |
| | | than the first injection – the last |
| | | injection hurt much less than the |
| | | first injection) |
| The DV3396 product hurt less | Dichotomous variable based on | Yes = "about the same" (includes |
| than or about the same as the | "Comparative pain experience" | "none of the products hurt loss |
| PDS290 product | variable above (Day 1) | "the DV3396 product hurt less |
| | | than the PDS290 product" or "the DV3396 product hurt much less |
| | | than the PDS290 product") |
| | | No = "The DV3396 product hurt |
| | | much more than the PDS290 |
| | | product" or "The DV3396 |
| | | product hurt more than the |
| | | PDS290 product" |

#### **Design and Treatments**

This is a single-center, cross-over, randomized, double-blind study in healthy men and women comparing the injection site <u>pain</u> experience of the DV3396 product to that of the PDS290 product when both products are used to deliver 0.25 mg semaglutide sc. Subjects will be randomized in a 2×2 scheme evenly to 4 sequences of product and injection side as in the table below:

| Treatment Short Identifier | Treatment Long Identifier | Ratio Required |
|---|---|---|
| First injection on right side, Second injection on left side | | |
| Α | DV3396 (Right) followed by PDS290 (Left) | 1 |
| С | PDS290 (Right) followed by DV3396 (Left) | 1 |
| First injection on left side, Second injection on right side | | |
| В | DV3396 (Left) followed by PDS290 (Right) | 1 |
| D | PDS290 (Left) followed by DV3396 (Right) | 1 |

Subjects will receive 2 single doses of semaglutide 0.25 mg on 1 day. The 2 products will be administered at least 30 minutes apart, in the anterior aspect of the abdominal wall on opposite sides of the midline.

An overview of the study design is given below:



#### Study Schedule

Screening : Between Day -21 and Day -1 Confinement period : One day in the clinic: Day 1

Follow-up : A follow-up phone call will take place between 4 and 5 weeks after drug

administration on Day 1

#### **Subjects**

A total of 104 subjects are planned to be randomized to achieve at least 100 completed subjects. The aim is to have an even distribution of male and female subjects in the study; at least 30% of the same sex should be randomized in the study.

#### **Key Inclusion Criteria**

- Male or female subjects, aged 18 to 75 years (both inclusive) at the time of signing informed consent.
- BMI ≥25.0 kg/m<sup>2</sup>
- Considered to be generally healthy based on the medical history, physical examination, and the results
  of vital signs, electrocardiogram (ECG), and clinical laboratory tests performed during the screening visit,
  as judged by the Investigator.

#### **Key Exclusion Criteria**

- Woman who is pregnant or breast-feeding or intends to become pregnant within 4 weeks after administration of the study drug, or is of childbearing potential and not using highly effective contraceptive methods with her fertile male sexual partner.
- Any disorder that in the Investigator's opinion might jeopardize subject's safety, evaluation of results, or compliance with the protocol.
- Glycosylated hemoglobin ≥6.5% at screening.
- Use of prescription medicinal products or non-prescription drugs or herbal products, except routine
  vitamins, topical medication, contraceptives, and occasional use of paracetamol (paracetamol not
  allowed within 24 hours prior to drug administration), within 14 days prior to drug administration.
- Average intake of more than 21 units of alcohol per week for male subjects and more than 14 units per week for female subjects: 1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits.
- Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at screening and admission to the clinical research center.
- Use of tobacco and nicotine products, defined as any of the below:
  - o Smoking more than 1 cigarette or the equivalent per day on average
  - Not able or willing to refrain from smoking and the use of nicotine substitute products during the in-house period
- Subject is not able to understand and read English or Dutch, or subject is not able to understand and comply with the study requirements.

#### Study Drug

| Material Number | Name | Name of Intervention Product |
|---|---|---|
| | Semaglutide B 1.34 mg/ml PDS290 | PDS290 product |
| | Semaglutide C 0.5 mg/ml DV3396 | DV3396 product |

#### **Variables**

Safety

: Intensity of injection site pain on a visual analogue scale (VAS), categorical assessment of injection site pain intensity (6-point scale), quality of pain modified SF-MPQ-2 inventory, duration of pain assessment, comparative pain assessment (5-point scale), adverse events, clinical laboratory (if postdose assessments are deemed relevant by the Investigator), physical examination (if postdose assessments are deemed relevant by the Investigator), 12-lead ECG (if postdose assessments are deemed relevant by the Investigator), and vital signs

#### **Statistical Methods**

Sample size calculation

: The sample size calculation considers both the primary endpoint and the dichotomous endpoints. Considering precision on the proportion of the dichotomous endpoints, a sample size of 100 subjects results in a confidence interval (CI) with a width of 10% on each side, eg, for a proportion of 60%, the CI is 60% (50%-70%).

A standard deviation of within-pair differences in VAS pain score between 2 subcutaneous injections was obtained from Novo Nordisk clinical trial INS-4011. The within-subject variance (adjusting for the effects of speed,

volume and injection region) was estimated to 348, corresponding to a standard deviation (SD) of the within-pair difference of  $\sqrt{(2\cdot348)}$  = 26 mm. A prospective study of acute pain found that the minimum clinically important difference for worsening of pain, ie, the difference on a VAS associated with the selection of "a little more pain" rather than "about the same" had a mean value of 10 mm.<sup>3</sup> With 100 subjects, a conservative standard deviation of 30 mm, and 90% power, it is possible to detect a difference smaller than 10 mm. Hence a sample size of 100 subjects is considered sufficient to detect a clinically important difference. Allowing for 4% dropouts or missing data, a total of 104 subjects will need to be randomized.

Analysis of endpoints

: The primary endpoint will be analyzed by a fixed analysis of variance model with VAS score as the dependent variable, and product, injection side (right side, left side), injection number (first injection, second injection), and subject as fixed effects. From the model, the difference in VAS score between the 2 products is estimated and presented with a 95% CI and a p-value. The interpretation of the difference in VAS pain scores will be supported and contextualized by the results of the analyses of the exploratory endpoints.

Descriptive statistics only will be applied for other safety parameters and secondary endpoints.

| Assessments | |
|-------------|-------|
| Schedule of | |
| Table 1 | Visit |

| Study Day | Days<br>-21 to -1 | ٥ | Day 1 | Day 29 to Day 36 |
|---|---|---|---|---|
| | | Predose | Dosing and After | |
| Ambulatory | × | × | × | × |
| Admission | | × | | |
| Discharge | | | × | |
| Informed Consent | × | | | |
| Medical History | × | | | |
| Previous Injection Experience <sup>a</sup> | × | | | |
| Demographics | × | | | |
| Physical Examination | × | | qΧ | |
| Body Height, Body Weight and BMI Calculation | × | | | |
| Serology (HBsAg, anti-HCV, anti-HIV-1 and -2) | × | | | |
| Urine Drug and Alcohol Screen | × | × | | |
| Urine Pregnancy Test (Females of Childbearing Potential Only) | × | × | | ×° |
| Clinical Laboratory <sup>d</sup> | × | | pΧ | |
| HbA1c HbA1c | × | | | |
| 12-lead ECG <sup>e</sup> | × | | ×e | |
| Vital Signs <sup>f</sup> | × | | × | |
| Eligibility Check | × | Xβ | | |
| Randomization and Stratification <sup>h</sup> | | × | | |
| Study Drug Administration <sup>h</sup> | | | × | |
| Intensity of Injection Site Pain VASi | | | × | |
| Categorical Assessment of Injection Site Pain Intensity | | | × | |
| Quality of Pain Modified SF-MPQ-2 Inventoryk | | | × | |
| Duration of Pain | | | × | |
| Comparative Pain Assessment <sup>m</sup> | | | × | |
| Previous and Concomitant Medication | × | × | × | × |
| AE Monitoring | × | × | × | × |
| Technical Complaints <sup>n</sup> | | × | × | |
| Drug Accountability | | | × | |

Physical examination: this will be a focused examination only done if deemed relevant by the Investigator

For the check on pregnancy at the follow-up phone call, female subjects of childbearing potential will be handed out a urine pregnancy test on Day 1. They will have to do the pregnancy test at the ealiest in the morning of Day 29 and at the latest in the morning of the follow-up phone call

The same tests may be done after the second study drug administration on Day 1 prior to discharge, if deemed relevant by the Investigator. Clinical laboratory tests (including clinical chemistry and hematology): at screening (non-fasting).

12-lead ECG may be done after the second study drug administration on Day 1 prior to discharge, if deemed relevant by the Investigator. 12-lead ECG: at screening.

Vital signs (supine systolic and diastolic blood pressure, and pulse): at screening and after the second study drug administration on Day 1 prior to discharge. Eligibility check on Day 1 before dosing concerns the urine pregnancy test (female subjects of childbearing potentialonly), urine drug and alcohol screen, and concomitant medication only.

Subjects will be randomized in a 2×2 scheme evenly to 4 sequences of product and injection side as in the table below:

| Ratio Required | le le | ~ | ~ | de | 1 | 1 |
|---|---|---|---|---|---|---|
| Treatment Long Identifier | First injection on right side, Second injection on left side | DV3396 (Right) followed by PDS290 (Left) | PDS290 (Right) followed by DV3396 (Left) | First injection on left side, Second injection on right side | DV3396 (Left) followed by PDS290 (Right) | PDS290 (Left) followed by DV3396 (Right) |
| Treatment Short Identifier | | ٧ | O | | В | Q |

Subjects will receive 2 single doses of semaglutide 0.25 mg on 1 day. The 2 products will be administered at least 30 minutes apart, in the anterior aspect of the abdominal wall on opposite sides of the midline

One minute after each injection, the VAS to rate the intensity of injection site pain will be administered.

The categorical assessment of injection site pain intensity (6-point scale) will be started after the VAS to rate the intensity of injection site pain has been completed after each injection.

The quality of pain modified SF-MPQ-2 inventory will be started after the categorical assessment of injection site pain intensity (6-point scale) has been completed after each injection.

Subjects have to indicate after each injection when the pain, if any, is gone.

The comparative pain assessment (5-point scale) comparing pain between the 2 injections will be completed after the second injection.

All technical complaints that occur, from the time of receipt of the product at the site until the time of the last usage of the product, must be collected and reported to Novo Nordisk.

# **TABLE OF CONTENTS**

| TIT | LE P | AGE | 1 |
|---|---|---|---|
| SP | ONS | OR AUTHORIZATION OF CLINICAL STUDY PROTOCOL | 2 |
| ΑU | | RIZATION OF CLINICAL STUDY PROTOCOL BY CONTRACT RESEAF | |
| СО | NTA | CT INFORMATION | 4 |
| SU | ММА | RY OF CHANGES | е |
| SYI | NOP | SIS | 7 |
| TAI | BLE | OF CONTENTS | 14 |
| TAI | BLE | OF TABLES | 16 |
| TAI | BLE | OF FIGURES | 17 |
| LIS | T OF | ABBREVIATIONS | 18 |
| 1. | INTE | RODUCTION | 19 |
| | 1.1 | Background | |
| | 1.2 | Risk-Benefit Assessment and Risk Mitigation | |
| | | 1.2.1 Anticipated Clinical Benefits | |
| | | 1.2.2 Risks Related to Semaglutide | |
| | | 1.2.3 Risks Associated with Participation in the Clinical Study | |
| | | 1.2.4 Possible Interactions with Concomitant Medical Treatments | 21 |
| | | 1.2.5 Risk Mitigation | 21 |
| | | 1.2.6 Risk-Benefit Rationale | 21 |
| | 1.3 | Study Rationale | 22 |
| 2. | OBJ | IECTIVES | 23 |
| 3. | END | POINTS | 23 |
| 4. | INVI | ESTIGATIONAL PLAN | 25 |
| | 4.1 | Overall Study Design and Plan | 25 |
| | | 4.1.1 Type of Study | 25 |

| | 4.1.2 | Screenin | g Period | | 25 |
|---|---|---|---|---|---|
| | 4.1.3 | Treatmer | nt Period | | 26 |
| | 4.1.4 | Follow-up | p | | 26 |
| 4.2 | Discu | ssion of S | Study Desig | n | 26 |
| 4.3 | Selec | tion of Stu | udy Populat | ion | 27 |
| | 4.3.1 | Inclusion | Criteria | | 27 |
| | 4.3.2 | Exclusion | n Criteria | | 27 |
| | 4.3.3 | Removal | of Subjects | from Assessment | 28 |
| 4.4 | Treatr | nents | | | 29 |
| | 4.4.1 | Treatmer | nts Administe | ered | 29 |
| | 4.4.2 | Identity o | of Investigation | onal Products | 29 |
| | 4.4.3 | | | Subjects to Treatment Groups | |
| | 4.4.4 | | | the Study | |
| | 4.4.5 | _ | | e Study | |
| | 4.4.6 | | | dy | |
| | 4.4.7 | _ | | | |
| | 4.4.8 | | | ion and Other Restrictions During the Study | |
| | | | | ce | |
| 4.5 | _ | | | Variables | |
| | 4.5.1 | • | | s Assessed and Schedule of Assessments | |
| | | 4.5.1.1 | • | Tolerability Measurements | |
| | | | 4.5.1.1.1<br>4.5.1.1.2 | Intensity of Injection Site Pain Visual Analogue Scale Categorical Assessment of Injection Site Pain Intensity. | |
| | | | 4.5.1.1.3 | Quality of Pain Modified SF-MPQ-2 Inventory | |
| | | | 4.5.1.1.4 | Duration of Pain | |
| | | | 4.5.1.1.5 | Comparative Pain Assessment (5-point scale) | |
| | | | 4.5.1.1.6<br>4.5.1.1.7 | Adverse Events Technical Complaints | |
| | | | 4.5.1.1.8 | Clinical Laboratory | |
| | | | 4.5.1.1.9 | Vital Signs | |
| | | | | Electrocardiogram | |
| | | 4512 | | Physical Examinationood Volume | |
| | 4.5.2 | 7.0.1.2 | | leasurements | |
| | 4.5.3 | | | odsdromons | |
| 4.6 | | • | | Determination of Sample Size | |
| 4.0 | 4.6.1 | | | Determination of Sample Size | |
| | 4.0.1 | 4.6.1.1 | | | |
| | | 4.6.1.2 | • | is set (FAS) | |
| | | 4.6.1.3 | | ol Set | |
| | 4.6.2 | | | ical Plan for Safety Evaluation | |
| | | 4.6.2.1 | • | of Safety and Tolerability | |
| | | | 4.6.2.1.1 | Intensity of Injection Site Pain Visual Analogue Scale | |
| | | | 4.6.2.1.2 | Categorical Assessment of Injection Site Pain Intensity,<br>Quality of Pain Modified SF-MPQ-2 Inventory, Duration | of |
| | | | 40040 | Pain, and Comparative Pain Assessment | |
| | | | 4.6.2.1.3 | Adverse Events | 45 |

| | | 4.6.2.1.4 Technical Complaints 4.6.2.1.5 Clinical Laboratory. 4.6.2.1.6 Vital Signs and Electrocardiograms 4.6.2.1.7 Physical Examination 4.6.3 Determination of Sample Size. 4.6.4 Interim Analysis | .45<br>.46<br>.46<br>.46 |
|---|---|---|---|
| | 4.7 | Data Quality Assurance | .46 |
| <b>5</b> . | ETH | IICS | . 48 |
| | 5.1 | Independent Ethics Committee | .48 |
| | 5.2 | Ethical Conduct of the Study | .48 |
| | 5.3 | Subject Information and Consent | .49 |
| | 5.4 | Privacy | .49 |
| 6 | etii | DY ADMINISTRATIVE STRUCTURE | 50 |
| 0. | 6.1 | Distribution of Activities | |
| | 6.2 | Documentation | |
| | 0.2 | 6.2.1 Archiving | |
| | | 6.2.2 Recording of Data in Source Documents and eCRFs | |
| _ | 001 | IEIDENTIALITY AND BURLICATION BOLLOY | |
| 7. | | NFIDENTIALITY AND PUBLICATION POLICY | |
| | 7.1<br>7.2 | Publication Policy | |
| | 1.2 | Dissemination of Clinical Trial Data | .52 |
| 8. | REF | ERENCES | . 53 |
| 9. | APP | PENDICES | . 54 |
| | 9.1 | Drug Accountability | .54 |
| | 9.2 | Adverse Events: Definitions and Procedures for Recording, Evaluation, Followand Reporting to Sponsor | _ |
| | | TABLE OF TABLES | |
| Tab | ole 1 | Schedule of Assessments | .12 |
| | ole 2 | Primary Endpoint | |
| | ole 3 | Exploratory Endpoints | |
| | ole 4 | Product and Side of Injection on Abdomen per Treatment | |
| | ole 6 | Visual Appearance and Function of the DV3396 Product and PDS290 Product | |
| | ole 7 | Number and Volume of Blood Samples and Total Blood Volume Collected per Subjection | |
| | ole 8 | Primary Endpoint. | |
| Tab | ole 9 | Exploratory Endpoints | |

| Table 10 | Detectable Difference with a Sample Size of 100 Subjects for Different Combinations of Power, and Standard Deviation | |
|---|---|---|
| | TABLE OF FIGURES | |
| Figure 1 | Overview of the Study Design | 5 |
| Figure 2 | Decision Tree for Determining the Event Type and the Respective Forms to | ) |
| | Complete with Associated Timelines 38 | 3 |

#### LIST OF ABBREVIATIONS

AE adverse event

ALAT (ALT) alanine aminotransferase ASAT (AST) aspartate aminotransferase

BMI body mass index CA Competent Authority

CHMP Committee for Medicinal Products for Human Use (formerly: Committee for

Proprietary Medicinal Products [CPMP])

CI confidence interval
CRF case report form
CSP clinical study protocol
CSR clinical study report
CTD Clinical Trial Directive

CV cardiovascular
DUN dispensing unit number
ECG electrocardiogram

eCRF electronic case report form
EDS Early Development Services
EMA European Medicines Agency

FAS full analysis set GCP Good Clinical Practice

GDPR General Data Protection Regulation

GI gastrointestinal
GLP glucagon-like peptide
HbA1c glycosylated hemoglobin
HBsAg hepatitis B surface antigen

HCV hepatitis C virus

HIV human immunodeficiency virus

IB investigator's brochure ICF informed consent form

ICH International Council for Harmonisation (formerly: International Conference on

Harmonisation)

IEC Independent Ethics Committee

MCID minimum clinically important difference

MEB Medicine Evaluation Board PCD primary completion date pharmacokinetic(s)

RA receptor agonist
SAE serious adverse event
SAP statistical analysis plan

sc subcutaneous SD standard deviation

SF-MPQ-2 Short-form McGill Pain Questionnaire 2

SOP standard operating procedure T2D type 2 diabetes mellitus

TEAE treatment-emergent adverse event

TMM trial materials manual
ULN upper limit of normal
VAS visual analogue scale
WMA World Medical Association

WMO Wet medisch-wetenschappelijk onderzoek met mensen (medical research

involving human subjects act)

#### 1. INTRODUCTION

#### 1.1 Background

Semaglutide is a potent glucagon-like peptide-1 (GLP-1) receptor agonist (RA) developed by Novo Nordisk for weight management (Project NN9536). Semaglutide has a half-life of approximately 160 hours, making it suitable for once-weekly dosing. Semaglutide is currently approved in the EU and other regions for 0.5 and 1 mg weekly subcutaneous (sc) administration for treatment of type 2 diabetes (T2D) (Ozempic). Weekly administration of semaglutide sc 2.4 mg is currently being evaluated in Phase 3a trials for weight management.

A 52-week Phase 2 dose-finding trial within weight management (NN9536-4153) has been completed. Relative to baseline, the estimated mean weight loss at week 52 was 13.8% at the highest dose tested (0.4 mg once-daily as an adjunct to diet and exercise) compared to the mean weight loss of 2.3% achieved by diet, exercise and placebo alone.

Clinical and nonclinical data indicate that the body weight-reducing effect of semaglutide is mainly mediated by a reduced energy intake. No unexpected safety findings were identified and the tolerability and safety profile were overall consistent with previous findings in the T2D development programme and the GLP-1 RA class in general.

The clinical development program for semaglutide sc was conducted with a cartridge-based prefilled PDS290 pen-injector.

For the weight management indication, Novo Nordisk is currently developing the DV3396 pen-injector, a single-dose pen-injector for sc injection of semaglutide, a new single-dose device with an integrated prefilled syringe.

The DV3396 pen-injector for the 0.25 mg dose (first escalation dose) houses a 1.0-mL syringe pre-filled with a 0.5-mL semaglutide solution. A semaglutide concentration of 0.5 mg/mL is used to obtain a dose of 0.25 mg. The device comes with a 29G regular-walled needle and is shield-activated, ie, the injection is activated when pushing the pen against the injection site.

To allow the DV3396 pen-injector to provide the semaglutide dose in a volume of 0.5 mL, a new semaglutide formulation has been required compared to the semaglutide formulation used for the PDS290 pen-injector. In addition to the change of semaglutide concentration, the preservative (phenol) is removed from the new formulation, as it is to be used for single injections, and the concentration of propylene glycol has been slightly increased to compensate for the absence of phenol and ensure isotonicity.

Detailed information about semaglutide sc, the PDS290 semaglutide pen-injector, and the DV3396 pen-injector are available in the investigator's brochure (IB).<sup>1</sup>

#### 1.2 Risk-Benefit Assessment and Risk Mitigation

#### 1.2.1 Anticipated Clinical Benefits

In the present study, healthy overweight/obese subjects are enrolled and they will therefore not benefit from the treatment with 2 single doses of semaglutide.

#### 1.2.2 Risks Related to Semaglutide

The sections below describe identified and potential risks associated with semaglutide treatment. For classification and further details of the risks, please refer to the IB.<sup>1</sup> The identified/potential risks are based on findings in nonclinical studies and clinical trials with semaglutide as well as with other GLP-1 RAs. For each of these risks, mitigating actions have been implemented to minimize the risks for subjects enrolled in this study.

#### Gastrointestinal adverse events

Consistent with findings with other GLP-1 RAs, the most frequently reported adverse events (AE) in clinical trials with semaglutide were gastrointestinal (GI) AEs. A low dose of semaglutide will be implemented in the study to mitigate the risk of GI AEs.

#### Cholelithiasis

Events of cholelithiasis were the most frequently reported gallbladder events in the Phase 2 weight management trial (NN9536-4153) and were in a few instances co-reported with the event adjudication committee confirmed acute pancreatitis. As a precaution, if cholelithiasis is suspected, appropriate clinical follow-up is to be initiated at the Investigator's discretion.

#### Acute pancreatitis

Acute pancreatitis has been observed with the use of GLP-1 RA drug class. As a precaution, subjects with a history of chronic pancreatitis or recent acute pancreatitis will not be enrolled in the study.

#### Medullary thyroid cancer (MTC)

Expected proliferative thyroid C-cell changes were seen in the mouse and rat carcinogenicity studies after daily exposure to semaglutide for 2 years. No hyperplasia was observed in monkeys after 52 weeks exposure up to 13-fold above the clinical plasma exposure at 2.4 mg/week. In clinical trials with semaglutide, there have been no clinically relevant changes in calcitonin levels. The C-cell changes in rodents are mediated by the GLP-1 receptor, which is not expressed in the normal human thyroid. Accordingly, the risk of GLP-1 receptor-mediated C-cell changes in humans is considered to be low. However, as a precaution, exclusion criteria related to medical history of multiple endocrine neoplasia type 2 are implemented in the study.

#### Pancreatic cancer

There is currently no support from nonclinical studies, clinical trials or postmarketing data that GLP-1 RA-based therapies increase the risk of pancreatic cancer, but pancreatic cancer has been classified as a potential class risk of GLP-1 RAs by the European

Medicines Agency (EMA). As a precaution, subjects with a history of malignant neoplasms within the past 5 years prior to screening will be excluded from the study.

#### Allergic reactions

As is the case with all protein-based pharmaceuticals, subjects treated with semaglutide are at risk of developing immunogenic and allergic reactions. As a precaution, subjects with known or suspected hypersensitivity to semaglutide or related products will not be enrolled in this study.

#### Pregnancy and fertility (based on nonclinical data)

Studies in animals have shown reproductive toxicity. There are limited data from the use of semaglutide in pregnant women. Therefore, semaglutide should not be used during pregnancy. Exclusion and discontinuation criteria related to pregnancy are implemented in the study.

#### 1.2.3 Risks Associated with Participation in the Clinical Study

In the current study, risks related with venous blood sampling are minimal as no PK samples will be collected; only a few blood samples will be taken for clinical laboratory evaluations.

#### 1.2.4 Possible Interactions with Concomitant Medical Treatments

Semaglutide delays gastric emptying and has the potential to impact the rate of absorption of concomitantly administered oral medicinal products. The potential effect of semaglutide on the absorption of co-administered oral medications was studied in trials at semaglutide 1 mg/week steady-state exposure. No clinically relevant drug-drug interactions with semaglutide were observed based on the evaluated medications.

#### 1.2.5 Risk Mitigation

All subjects in this study will have a thorough medical check before entering the study. During the study, they will be followed closely and carefully by qualified medical staff. This will mitigate the known and potential risks.

#### 1.2.6 Risk-Benefit Rationale

The healthy subjects enrolled in the study will not have immediate health benefits from participating in this study. Data from this study might, however, benefit future treatment of subjects with T2D and overweight/obesity through a more convenient drug administration with the DV3396 product than with the PDS290 semaglutide product. The safety profile of semaglutide is well documented; AEs were mostly predictable based on the known effects of GLP-1 RAs. Thus, based on the large nonclinical and clinical development program with semaglutide 1.34 mg/mL and on the usability evaluation of the DV3396 product, it is concluded that there are no safety issues that would prohibit administration of semaglutide in accordance with the planned clinical study.

More detailed information about the known and expected benefits and risks and reasonably expected AEs of semaglutide sc, the PDS290 semaglutide pen-injector, and the DV3396 pen-injector are available in the IB.<sup>1</sup>

#### 1.3 Study Rationale

Novo Nordisk is currently developing the DV3396 pen-injector for the sc administration of semaglutide, the drug that is currently marketed for T2D in the PDS290 pen-injector in a different formulation. To evaluate the injection site *pain* experience after a single dose of semaglutide sc 0.25 mg, the present explorative study compares injection pain between the DV3396 product and the PDS290 pen-injector used with the Ypsomed Clickfine AutoProtect, 8 mm x 29G needle: The Ypsomed Clickfine® AutoProtect, 8 mm x 29G needle is chosen for its similarity to the built-in needle of the DV3396 product and is larger than the needle with which the PDS290 pen-injector is commercialized. Together, the PDS290 pen-injector and the Ypsomed Clickfine® AutoProtect, 8 mm x 29G needle will be referred to as the PDS290 product.

#### 2. OBJECTIVES

The primary objective is to compare, in healthy subjects, the injection site  $\underline{pain}$  experience of a single dose of 0.25 mg semaglutide sc, given as the DV3396 product to that of the PDS290 product.

# 3. ENDPOINTS

**Table 2** Primary Endpoint

| Endpoint Title | Time Frame | Unit |
|---|---|---|
| Intensity of injection site pain | 1 min after each injection (Day 1) | mm on a 100-mm horizontal visual analogue scale |
| | | (where 0 mm = no pain, |
| | | 100 mm = unbearable pain) |

**Table 3** Exploratory Endpoints

| Endpoint Title | Time Frame | Unit |
|---|---|---|
| Categorical assessment of injection site pain intensity | Immediately after rating of intensity of injection site pain, | 6-point scale (none – very mild – mild – moderate – severe – |
| anyonon one pain anotony | ie, after 1 min plus the time it<br>takes to complete the rating of<br>intensity of injection site pain by | very severe) |
| Moderate or more injection site pain | visual analogue scale (Day 1) Dichotomous variable based on categorical assessment of | Yes = moderate, severe, very severe |
| | intensity of injection site pain (Day 1) (item above) | No = none, very mild, mild |
| Quality of pain | Immediately after categorical assessment of intensity of injection site pain, ie, after 1 | Pain quality items on modified SF-MPQ-2 inventory (select all that apply): |
| | min plus the time it takes to complete the rating of intensity | Throbbing pain □ |
| | of injection site pain and the | Shooting pain □ |
| | categorical rating of intensity of | Stabbing pain □<br>Sharp pain □ |
| | injection site pain (Day 1) | Cramping pain □ |
| | | Gnawing pain □ |
| | | Hot-burning pain □ |
| | | Aching pain □ |
| | | Heavy pain □ |
| | | Tender □ |
| | | Splitting pain □ |
| | | Tiring-exhausting □ |
| | | Sickening □ |
| | | Fearful □ |
| | | Punishing-cruel □ |
| | | Electric-shock pain □ |
| | | Cold-freezing pain □ |
| Duration of nain | From time of injection : | Piercing |
| Duration of pain | From time of injection until cessation of pain (Day 1) | min and sec |

| Endpoint Title | Time Frame | Unit |
|---|---|---|
| Comparative pain experience | After pain has ended after the | 5-point scale (the last injection |
| | last injection (Day 1) | hurt much more than the first |
| | | injection – the last injection hurt |
| | | more than the first injection - |
| | | they hurt about the same |
| | | [includes: none of the injections |
| | | hurt] – the last injection hurt |
| | | less than the first injection – the |
| | | last injection hurt much less |
| | | than the first injection) |
| The DV3396 product hurt less | Dichotomous variable based | Yes = "about the same" |
| than or about the same as the | on "Comparative pain | (includes "none of the products |
| PDS290 product | experience" variable above | hurt" or "the DV3396 product |
| | (Day 1) | hurt less than the PDS290 |
| | | product" or "the DV3396 |
| | | product hurt much less than the |
| | | PDS290 product") |
| | | No = "The DV3396 product hurt |
| | | much more than the PDS290 |
| | | product" or "The DV3396 |
| | | product hurt more than the |
| | | PDS290 product" |

#### 4. INVESTIGATIONAL PLAN

#### 4.1 Overall Study Design and Plan

#### 4.1.1 Type of Study

This is a single-center, cross-over, randomized, double-blind study in healthy men and women comparing the injection site <u>pain</u> experience of the DV3396 product to that of the PDS290 product when both products are used to deliver 0.25 mg semaglutide sc. Subjects will be randomized in a 2×2 scheme evenly to 4 sequences of product and injection side as in Table 4.

Table 4 Product and Side of Injection on Abdomen per Treatment

| Treatment<br>Short Identifier | Treatment Long Identifier | Ratio Required |
|---|---|---|
| First injection on right side, Second injection on left side | | |
| A | DV3396 (Right) followed by PDS290 (Left) | 1 |
| С | PDS290 (Right) followed by DV3396 (Left) | 1 |
| | First injection on left side, Second injection on right side | |
| В | DV3396 (Left) followed by PDS290 (Right) | 1 |
| D | PDS290 (Left) followed by DV3396 (Right) | 1 |

Subjects will receive 2 single doses of semaglutide 0.25 mg on 1 day. The 2 products will be administered at least 30 minutes apart, in the anterior aspect of the abdominal wall on opposite sides of the midline.

The end of the study is defined as last subject last visit (last follow-up phone contact).

An overview of the study design is given in Figure 1.

Figure 1 Overview of the Study Design



#### 4.1.2 Screening Period

Subjects will report to the medical screening facility for the eligibility screening (see Section 4.3 for inclusion and exclusion criteria) within 3 weeks prior to drug administration.

Subjects will sign the study-specific informed consent form (ICF) prior to any study-specific screening procedures being performed. The written informed consent will be obtained for all subjects, regardless of their eligibility for the study; the signed ICFs will be retained and archived at to the subject.

Eligibility screening will consist of the assessments as presented in the schedule of assessments (Table 1).

#### 4.1.3 Treatment Period

Subjects will be in the clinic research center for 1 day, on Day 1. On this day, the subjects will be admitted, the drug will be administered twice, and the subjects will be discharged after all assessments have been performed.

If the subject admits to bodily pain (eg, headache) at admission (Day 1), then Day 1 should be rescheduled within the visit window as the existing pain could impact the injection pain assessment.

Assessments during the treatment period will be performed as presented in the schedule of assessments (Table 1).

#### 4.1.4 Follow-up

A follow-up phone call will take place between 4 and 5 weeks after drug administration on Day 1.

#### 4.2 Discussion of Study Design

A total of 104 subjects are planned to be randomized to achieve at least 100 completed subjects. The aim is to have an even distribution of males and females in the study; at least 30% of the same sex should be randomized in the study.

Subjects with a body mass index (BMI) ≥25.0 kg/m² but generally healthy will be included to minimize inter-subject variability due to frequent comorbidities in the target users of semaglutide (T2D and general population with overweight/obesity). It is assumed that the ability to detect differences between the 2 formulations does not differ between healthy subjects and target users. Only subjects with a BMI greater than or equal to 25 kg/m² will be included to reduce the risk of intramuscular injection. Both male and female subjects will be included to ensure generalizability to the intended users of both genders. Only individuals of age 18 years or older are eligible because semaglutide sc is only approved for use in adults with T2D. The upper age limit of 75 years is justified by the cognitive demands of the subjects when completing the inventories used in this study.

The length of the cross-over interval is set to be as short as possible to minimize systemic effects of semaglutide, especially nausea, between the first and the last injection, while being long enough to minimize residual pain and emotional carry-over from the first injection.

#### 4.3 Selection of Study Population

#### 4.3.1 Inclusion Criteria

Note: Restrictions that apply to the period after admission are described in Section 4.4.8, except when they concern a statement of willingness.

The following inclusion criteria must be met for a subject to be eligible for inclusion in the study:

- Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
- 2. Male or female subjects, aged 18 to 75 years (both inclusive) at the time of signing informed consent.
- 3. BMI ≥25.0 kg/m<sup>2</sup>
- 4. Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram, and clinical laboratory tests performed during the screening visit, as judged by the Investigator.

#### 4.3.2 Exclusion Criteria

Note: Restrictions that apply to the period after admission are described in Section 4.4.8, except when they concern a statement of willingness.

A subject who meets any of the following exclusion criteria will not be eligible for inclusion in the study:

- 1. Known or suspected hypersensitivity to the study product or related products.
- 2. Previous participation in this study. Participation is defined as having received investigational product.
- 3. Woman who is pregnant or breast-feeding or intends to become pregnant within 4 weeks after administration of the study drug, or is of childbearing potential and not using highly effective contraceptive methods with her fertile male sexual partner (see Section 4.4.8 for details on highly effective contraception).
- 4. Participation in a drug study within 60 days prior to drug administration in the current study. Participation in more than 4 other drug studies in the 12 months prior to drug administration in the current study.
- 5. Any disorder that in the Investigator's opinion might jeopardize subject's safety, evaluation of results, or compliance with the protocol.
- 6. Glycosylated hemoglobin (HbA1c) ≥6.5% at screening.
- 7. Supine blood pressure at screening (after resting for at least 5 minutes) outside the range of 90 to 160 mmHg for systolic or 45 to 89 mmHg for diastolic.
- 8. Supine pulse rate (as part of vital signs) (after resting for at least 5 minutes) outside the range of 40 to 100 beats per minute.
- 9. Use of prescription medicinal products or non-prescription drugs or herbal products, except routine vitamins, topical medication, contraceptives, and occasional use of paracetamol (paracetamol not allowed within 24 hours prior to drug administration), within 14 days prior to drug administration.

- 10. Diagnostic test results positive for human immunodeficiency virus (HIV)-1 or HIV-2 infection.
- 11. Diagnostic test results positive for hepatitis B or hepatitis C infection.
- 12. Mental incapacity, language barriers, or unwillingness to comply with the requirements of the protocol, which may preclude adequate understanding or cooperation during the study as judged by the Investigator.
- 13. Average intake of more than 21 units of alcohol per week for male subjects and more than 14 units per week for female subjects: 1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits.
- 14. Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at screening and admission to the clinical research center.
- 15. Use of tobacco and nicotine products, defined as any of the below:
  - Smoking more than 1 cigarette or the equivalent per day on average
  - Not able or willing to refrain from smoking and the use of nicotine substitute products during the in-house period
- 16. Blood donation, plasma donation or blood draw (as declared by the subject or reported in the medical records):
  - In excess of 400 mL within the past 90 days prior to the day of screening
  - In excess of 50 mL within the past 30 days prior to the day of screening
- Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma (as declared by the subject or reported in the medical records)
- 18. Subjects with a history of malignant neoplasms within the past 5 years prior to screening.
- 19. Presence or history of pancreatitis (acute or chronic; as declared by the subject or reported in the medical records).
- 20. Subject is not able to understand and read English or Dutch, or subject is not able to understand and comply with the study requirements.
- 21. Subject depends on the Sponsor, the Investigator, or the study center, or subject is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the study.
- 22. Vulnerable subject (eg, person kept in detention) who may have an increased likelihood of being wronged or of incurring additional harm.

Please note that subjects should refrain from consumption of any foods containing poppy seeds and alcohol within 48 hours (2 days) prior to screening and admission to the clinical research center to avoid false-positive drug screen results. In addition, they should refrain from strenuous exercise within 96 hours (4 days) prior to screening and admission as this could result in abnormal clinical laboratory values.

#### 4.3.3 Removal of Subjects from Assessment

Participation in the study is strictly voluntary. A subject has the right to withdraw from the study at any time for any reason.

The subject may be discontinued at any time during the study at the discretion of the Investigator for safety, behavioral, compliance, or administrative reasons.

If a subject is withdrawn from the study, the Sponsor will be informed immediately. If there is a medical reason for withdrawal, the subject will remain under the supervision of the Investigator until satisfactory health has returned.

Subjects who drop out or withdraw for any reason without completing all screening evaluations successfully will be considered screening failures.

A subject who is withdrawn or voluntarily withdraws from the study for any reason, whether related to the study product or not, after having received a subject number, will be considered an early-termination subject. Early-termination subjects will not be replaced.

will make every effort to ensure that early-termination subjects who have received study drug complete the safety follow-up assessments.

#### 4.4 Treatments

#### 4.4.1 Treatments Administered

Subjects will be randomized in a 2×2 scheme evenly to 4 sequences of product and injection side as in Table 4 in Section 4.1.1. Subjects will receive 2 single doses of semaglutide 0.25 mg on 1 day. The 2 products will be administered at least 30 minutes apart, in the anterior aspect of the abdominal wall on opposite sides of the midline.

Unblinded members of the staff not otherwise involved in the study procedures will be responsible for study drug administration. In each subject, the 2 semaglutide injections should be performed by the same staff member.

The staff member will be instructed to select an injection site on the assigned side of the midline, that, according to their judgment based on visual inspection and palpation, has the maximal thickness of subcutaneous fat. The injection with the DV3396 product will be performed as described in the DV3396 pen-injector directions for use, ie, without making a lifted skin fold. Injection with the PDS290 product will be performed as described in the PDS290 pen-injector directions for use and the Ypsomed Clickfine AutoProtect, 8 mm x 29G needle instructions for use. However, to standardize the injections, using a lifted skin fold with the PDS290 product will not be an option.

The unblinded staff will instruct the subject to avoid discussing the administration of the study drug with other study staff including the Investigator.

#### 4.4.2 Identity of Investigational Products

Novo Nordisk A/S Denmark will supply the following products:

Table 5 Products Supplied by Novo Nordisk A/S

| Material Number | Name | Name of Intervention Product |
|---|---|---|
| | Semaglutide B 1.34 mg/ml PDS290 | PDS290 product |
| | Semaglutide C 0.5 mg/ml DV3396 | DV3396 product |

In this study only, the PDS290 product will be used with an Ypsomed Clickfine AutoProtect, 8 mm x 29G needle. This needle will be sourced directly by

For details concerning drug storage and drug accountability see Appendix 9.1.

The characteristics of the 2 products are shown in Table 6.

Table 6 Visual Appearance and Function of the DV3396 Product and PDS290 Product

| 110000 | | |
|---|---|---|
| | DV3396 product | PDS290 product |
| Appearance (colours and labelling not final) | | |
| Uses | Single | Multiple |
| Length (with cap) | 123 mm | 138 mm |
| Diameter | 17 mm | 19 mm |
| Housing colour | White | Light blue |
| Dose volume (0.25 mg) | 0.5 mL | 0.19 mL |
| Needle | Integrated and hidden, 6 mm, 29 G | Must be attached before injection: Ypsomed Clickfine® AutoProtect, 8 mm x 29G* |
| Activation mechanism | Needle shield | Dose button |

<sup>\*</sup> Needle used with the PDS290 product is specific to study INS-4582

All dose administrations will be performed by trained, unblinded staff at the study site.

Directions for use of all products provided by Novo Nordisk are provided in the Trial Materials Manual (TMM) also provided by Novo Nordisk.

#### 4.4.3 Method of Assigning Subjects to Treatment Groups

After obtaining informed consent, subjects will be screened according to the inclusion and exclusion criteria. Subjects who have met all eligibility criteria will receive a subject number upon inclusion in the study. They receive the subject number just prior to dosing. The subject number will ensure identification throughout the study.

The subject number will be the same as the randomization number given on the randomization list produced by Novo Nordisk. The randomization list will be transferred to the Pharmacy and kept in a restricted area to which only the Pharmacy has access.

Subjects will be randomized in a 2×2 scheme evenly to 4 sequences of product and injection side as described in Section 4.1.1. Subjects will receive a randomization

number based on the randomization list produced by Novo Nordisk. The randomization number encodes the assignment to one of the 4 sequences. The randomization list will be transferred to the Pharmacy and kept in a restricted area to which only the Pharmacy has access.

Subjects who drop out or withdraw for any reason without completing all screening evaluations successfully will be considered screening failures. Such subjects, and also subjects who are eligible for inclusion in the study but do not receive the study drug, will not receive a subject number, and only applicable data will be entered in the electronic case report forms (eCRFs).

#### 4.4.4 Selection of Doses in the Study

The lowest available dose for DV3396 product is 0.25 mg. Hence, to compare the DV3396 and PDS290 products, a dose of 0.25 mg has been chosen for both products. The subject will receive 2 injections at least 30 minutes apart giving a total dose of 0.5 mg, which is the highest single dose of semaglutide tolerated without dose escalation due to risk of GI AEs.

#### 4.4.5 Timing of Doses in the Study

The first dose will be administered as follows. A blinded staff member who is present in the study room will start a timer when the unblinded staff member starts the injection. The timer will be placed such that it is not visible to the subject. The subject will be instructed to indicate when all pain is gone. If no pain is experienced, "00 min, 00 s (sec)" will be recorded.

One minute after the injection, the blinded staff member will administer the visual analogue scale (VAS) to rate the intensity of injection site pain (not the momentary pain at the time of VAS completion) (see Section 4.5.1.1.1).

When the subject has completed the intensity of injection site pain VAS after the first injection of the study drug, the subject will complete a categorical assessment of injection site pain intensity (6-point scale) (see Section 4.5.1.1.2) and then a quality of pain modified SF-MPQ-2 inventory (see Section 4.5.1.1.3).

Because the completion of the inventories may distract the subject, they will be reminded at regular intervals to indicate when the pain, if any, is gone, if they have not already done so.

At least 30 minutes after the first injection, after confirmation from the subject that the pain is entirely gone (to not contaminate the rating of the last injection), the timer will be reset, and the last injection will be given. If the pain is not gone at 30 minutes, another attempt will be made at 60 minutes. If pain is still present at that time, no further attempts will be made.

Following the last injection, the same measurements will be performed as after the first injection, as described above. Subjects will not be allowed to consult their own prior

ratings. After confirmation from the subject that the pain is entirely gone, the subjects will complete a comparative pain assessment (5-point scale) comparing pain between injections (see Section 4.5.1.1.4).

During the 30 minutes after each administration of the study drug the subjects should stay in bed or should be seated in a chair, and not walk around.

#### 4.4.6 Meals During the Study

There are no requirements with regard to fed or fasting conditions prior to or after study drug administration. Further, no fasting is required before obtaining clinical laboratory samples.

With the exception of the restrictions with respect to methylxanthine- and alcohol-containing beverages or food, as described in Section 4.4.8, there are no special requirements related to food and beverage intake. Meals and snacks (such as decaffeinated coffee, herbal tea, fruit, biscuits) will be provided according to standard operating procedures (SOPs).

#### 4.4.7 Blinding

This is a double-blind study.

Investigators will remain blinded to each subject's assigned product throughout the course of the study. Also, all staff not participating in unblinded tasks will be blinded to treatment. To maintain this blind, qualified, unblinded members of the staff not otherwise involved in the study procedures will be responsible for study drug administration according to the randomization list. Technical complaints will also be collected by unblinded site staff. The unblinded staff will not be involved in any other assessments or safety reporting.

Subjects will be blinded to treatment as well. To maintain blinding of subjects, a visual blind will be in place during dose administration. To maintain blinding of staff present in the room during administration (for timekeeping, etc.), an acoustic blind will be in place (eg, headphones or white noise).

The randomization list will be provided to the pharmacist at for dispensing purposes and kept in the pharmacy, accessible to the pharmacist, the pharmacy assistant, and the unblinded staff only.

Individual code break envelopes will be provided for all subjects by Novo Nordisk. Each sealed envelope containing the sequence will be kept in a medication storage room, which is locked with restricted access. To manage the subject's condition in case of a medical emergency, the Investigator is allowed to break the code to know which semaglutide formulation was administered (using which product). The date when and reason why the blind was broken must be recorded in the source documentation. The Sponsor (Global Safety department) and unblinded monitor will be informed in case of unblinding.

#### 4.4.8 Concomitant Medication and Other Restrictions During the Study

Note: Restrictions that apply to the period before admission are described in Section 4.3.1 and Section 4.3.2.

The use of all prescription medicinal products or non-prescription drugs or herbal products is not allowed from admission to the clinical research center until discharge. An exception is made for routine vitamins, topical medication, and contraceptives, which are allowed throughout the study. During the stay in the clinical research center, the Investigator may permit a limited amount of paracetamol for the treatment of headache or any other pain, but this is only allowed after all pain assessments have been completed. Other medication to treat AEs during the stay in the clinical research center may only be prescribed if deemed necessary by the Investigator. If medication is used during the stay in the clinical research center, the name of the drug, the dose, and dosage regimen will be recorded in the eCRF. Any medication taken between discharge and the follow-up phone call will be documented in a similar fashion.

The use of alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks), grapefruit (juice), and tobacco products is not allowed during the stay in the clinical research center.

Strenuous exercise is not allowed during the stay in the clinical research center.

No contraception measures are required for male subjects as the risk of teratogenicity/fetotoxicity caused by transfer of semaglutide in seminal fluid is unlikely.

Female subjects of childbearing potential who have a fertile male sexual partner must agree to use highly effective contraception from screening up to 4 weeks after drug administration. Highly effective contraception is defined as:

- Use of combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal [patch]), or
- Use of progestogen-only hormonal contraception associated with inhibition of ovulation (oral or injectable).

The above requirements on contraception do not apply if:

- The male partner of the female subject is vasectomized and has a confirmed post-vasectomy semen analysis.
- The female subject practices sexual abstinence during the period mentioned above.

#### 4.4.9 Treatment Compliance

Each of the single doses will be administered by trained unblinded staff at the clinical research center. The exact times of study drug administration will be recorded in the eCRF.

#### 4.5 Safety Measurements and Variables

Only safety parameters will be assessed in this study; the study does not comprise efficacy, pharmacokinetic, or pharmacodynamic measurements.

#### 4.5.1 Safety Measurements Assessed and Schedule of Assessments

A schedule of assessments is presented in Table 1.

#### 4.5.1.1 Safety and Tolerability Measurements

Safety and tolerability assessments will consist of intensity of injection site pain VAS, categorical assessment of injection site pain intensity (6-point scale), quality of pain modified SF-MPQ-2 inventory, duration of pain assessment, comparative pain assessment (5-point scale), AEs, clinical laboratory, vital signs, and 12-lead electrocardiogram (ECG). In addition, some assessments will only be performed at screening or predose for the assessment of eligibility and are also described in this section.

All assessments will be performed in accordance with the schedule of assessments (Table 1).

#### 4.5.1.1.1 Intensity of Injection Site Pain Visual Analogue Scale

The intensity of injection site pain VAS will be filled in by the subjects starting 1 minute after each injection of the study drug to report the pain intensity experienced in the first minute after the injection.

Subjects will be instructed to make a vertical line on the VAS (100 mm); the endpoints are "no pain" and "unbearable pain." The distance (mm) between the endpoint "no pain" and the vertical line on the VAS will be recorded in the eCRF.

#### First injection

English version:

Indicate the intensity of pain you felt during the injection. For this, make a vertical line somewhere through the line below, where the endpoints are "no pain" and "unbearable pain".



#### Last injection

English version:

Indicate the intensity of pain you felt during the last injection only. For this, make a vertical line somewhere through the line below, where the endpoints are "no pain" and "unbearable pain".


## 4.5.1.1.2 Categorical Assessment of Injection Site Pain Intensity

The categorical assessment of injection site pain intensity is a 6-point scale in which the pain intensity is rated by the subjects as follows:

Please tick one box describing the pain intensity during the injection:

| none |
|-------------|
| very mild |
| mild |
| moderate |
| severe |
| very severe |

Please tick one box describing the pain intensity during the last injection only:

| none |
|-------------|
| very mild |
| mild |
| moderate |
| severe |
| very severe |

## 4.5.1.1.3 Quality of Pain Modified SF-MPQ-2 Inventory

The quality of pain will be assessed using the modified short-form McGill pain questionnaire (modified SF-MPQ-2 inventory<sup>2</sup>) to be filled in by the subjects as follows:

This questionnaire provides you with a list of words that describe some of the different qualities of pain and related symptoms. Please put an X in all boxes that apply:

| Throbbing pain |
|---------------------|
| Shooting pain |
| Stabbing pain |
| Sharp pain |
| Cramping pain |
| Gnawing pain |
| Hot-burning pain |
| Aching pain |
| Heavy pain |
| Tender |
| Splitting pain |
| Tiring-exhausting |
| Sickening |
| Fearful |
| Punishing-cruel |
| Electric-shock pain |
| Cold-freezing pain |
| Piercing |

#### 4.5.1.1.4 Duration of Pain

The duration of pain as indicated by the subject will be recorded from time of injection until cessation of pain in minutes and seconds.

## 4.5.1.1.5 Comparative Pain Assessment (5-point scale)

The comparative pain assessment is a 5-point scale in which the subjects will compared the pain between the 2 injections.

## The subjects will be asked to answer the following question:

Please choose the statement below that best describes your experience:

- The last injection hurt much more than the first injection.
- The last injection hurt more than the first injection.
- They hurt about the same (includes: none of the injections hurt).
- The last injection hurt less than the first injection.
- The last injection hurt much less than the first injection.

#### 4.5.1.1.6 Adverse Events

The definitions of AEs and serious AEs (SAEs) can be found in Appendix 9.2.

The Investigator is responsible for detecting, documenting, recording, and following up on events that meet the definition of an AE or SAE.

## Time period and frequency for collecting AE and SAE information

All AEs will be collected from the first study-related activity after obtaining informed consent and until the follow-up visit at the time points specified in the schedule of assessments (Table 1).

All SAEs will be recorded and reported to Novo Nordisk or designee within 24 hours, as indicated in Appendix 9.2. The investigator must submit any updated SAE data to Novo Nordisk within 24 hours of it being available.

Investigators are not obligated to actively seek AEs or SAEs in former study subjects. However, if the Investigator learns of any SAE, including a death, at any time after a subject has been discontinued from/completed the study, and the Investigator considers the event to be possibly/probably related to the investigational study product or study participation, the investigator must promptly notify Novo Nordisk.

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 9.2.

Timelines for reporting of AEs are listed in Figure 2.

Medication error AEs require additional data collection via a specific event form. For definition of medication errors, see Appendix 9.2.

In order for Novo Nordisk to perform a complete investigation of reported SAEs, Novo Nordisk might ask the Investigator to complete a technical complaint form. For reporting of technical complaints, see Section 4.5.1.1.7.

The reporting timelines are specified in Figure 2.

Figure 2 Decision Tree for Determining the Event Type and the Respective Forms to Complete with Associated Timelines



#### Method of detecting AEs and SAEs

Care should be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the subject is the preferred method to inquire about events.

#### Follow-up on AEs and SAEs

After the initial AE/SAE report, the Investigator is required to proactively follow each subject at subsequent visits/contacts. All SAEs will be followed until resolution, stabilization, or if the event is otherwise explained (eg, chronic condition), or the subject is lost to follow-up. Further information on follow-up procedures is given in Appendix 9.2.

### Regulatory reporting requirements for SAEs

Prompt notification by the Investigator to Novo Nordisk of an SAE (according to Figure 2 and Appendix 9.2) is essential so that legal obligations and ethical responsibilities towards the safety of subjects and the safety of a study product under clinical investigation are met.

Novo Nordisk has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study product under clinical investigation. Novo Nordisk will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, the Independent Ethics Committee (IEC), and investigators.

Safety reports must be prepared for suspected unexpected serious adverse reactions according to local regulatory requirements and Novo Nordisk policy and forwarded to regulatory authorities, IEC, and investigators as locally required.

An Investigator who receives an investigator safety report describing a SAE or other specific safety information (eg, summary or listing of SAEs), from Novo Nordisk will review and then file it along with the IB and will notify the IEC, if appropriate, according to local requirements.

#### Pregnancies and associated adverse events

Details of pregnancies in female subjects will be collected after the first study-related activity after obtaining informed consent and until pregnancy outcome.

If a pregnancy is reported in a female subject, the investigator should inform Novo Nordisk within 14 calendar days of learning of the pregnancy and should follow the procedures outlined below:

- The Investigator will collect pregnancy information on any female subject, who becomes pregnant while participating in this study.
- Information will be recorded on the appropriate form and submitted to Novo Nordisk within 14 calendar days of learning of a subject's pregnancy.
- Subject will be followed to determine the outcome of the pregnancy. The Investigator
  will collect follow-up information on the subject and neonate, which will be forwarded
  to Novo Nordisk. Generally, follow-up will not be required for longer than 1 month
  beyond the delivery date.
- Any termination of pregnancy will be reported, regardless of fetal status (presence or absence of anomalies) or indication for procedure.
- Although pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy will be reported as an AE or SAE.
- A spontaneous abortion is always considered to be an SAE and will be reported as such.
- Any SAE occurring as a result of a post-study pregnancy that is considered
  possibly/probably related to the study product by the Investigator will be reported to
  Novo Nordisk as described in Appendix 9.2. Although the Investigator is not
  obligated to actively seek this information in former subjects, he or she may learn of
  an SAE through spontaneous reporting.

Any female subject who becomes pregnant while participating in the study will discontinue study product.

Pregnancy outcome should be documented in the subject's medical record. An abnormal pregnancy outcome (eg, spontaneous abortion, fetal death, stillbirth, congenital anomaly, and ectopic pregnancy) is considered an SAE.

### 4.5.1.1.7 Technical Complaints

The unblinded staff is responsible for the detection and documentation of technical complaints that occur when using the pen-injectors used in this study.

#### Definition of technical complaint:

 A technical complaint is any written, electronic or oral communication that alleges medical product defects and device product defects. The technical complaint may be associated with an AE, but does not concern the AE itself.

Examples of technical complaints are as follows:

- Problems with the physical or chemical appearance of study products (eg, discoloration, particles or contamination).
- Problems with packaging material including labelling.
- Problems related to pen-injectors (eg, to the injection mechanism, dose setting mechanism, push button, or interface between the pen-injector and the needle).

The Investigator must assess whether a technical complaint is related to an AE.

## Time period for detecting technical complaints

All technical complaints that occur from the time of receipt of the product at until the time of the last usage of the product must be collected for products predefined on the technical complaint form.

### Reporting of technical complaints to Novo Nordisk

Technical complaints must be reported on a separate technical complaint form:

- One technical complaint form must be completed for each affected dispensing unit number (DUN).
- If a DUN is not available, a technical complaint form for each batch, code, or lot number must be completed.

#### Timelines for reporting of technical complaints to Novo Nordisk

The Investigator must complete as much information on the form as possible and hand it over to the unblinded staff. The unblinded staff must fill in the unblinded information on the form (such as the DUN and batch, code, or lot number) and forward the technical complaint form to the Customer Complaint Center, Novo Nordisk, within the timelines specified below:

- Technical complaints related to SAEs, within 24 hours
- All other technical complaints, within 5 calendar days

The technical complaint form must be kept inaccessible for blinded site staff.

#### Follow-up of technical complaints

The Investigator is responsible for ensuring that new or updated information will be recorded on the originally completed form.



The unblinded staff must collect the technical complaint sample and all associated parts that were packed in same DUN. The unblinded staff collects the sample and

notify the unblinded monitor within 5 calendar days of obtaining the sample at The sample and all associated parts must be sent as soon as possible to Customer Complaint Center, Novo Nordisk, together with a copy of the completed technical complaint form.

The technical complaint sample should contain the batch, code, or lot number and, if available, the DUN. If the technical complaint sample is unobtainable, the reason must be stated on the technical compliant form.

If several samples are shipped in one shipment, the sample and the corresponding technical complaint form should be kept together.

Storage for the technical complaint sample must be done in accordance with the conditions prescribed for the product.

# Reporting of technical complaints for Novo Nordisk products not included in technical complaint form

Technical complaints on Novo Nordisk products not included in the technical complaint form should be reported to local Novo Nordisk affiliate with a reference to trial ID.

### 4.5.1.1.8 Clinical Laboratory

Blood and urine samples for clinical laboratory assessments will be collected according to SOPs. No fasting is required prior to collecting these samples.

The following parameters will be measured:

- Clinical chemistry (serum quantitatively): total bilirubin, alkaline phosphatase, aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), creatinine, albumin, sodium, potassium, and calcium.
- Hematology (blood quantitatively): leukocytes, hemoglobin, and thrombocytes. HbA1c at screening only.
- Serology:

hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), and anti-human immunodeficiency virus (HIV)-1 and -2.

- Drug and alcohol screen:
   opiates, methadone, cocaine, amphetamines (including ecstasy), cannabinoids,
   barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol in urine.
- Hormones (serum quantitatively): thyroid-stimulating hormone.
- Pregnancy test (female subjects of childbearing potential only):
   β-human chorionic gonadotropin in urine.

In case of unexplained or unexpected clinical laboratory test values, the tests will be repeated as soon as possible and followed up until the results have returned to the normal range and/or an adequate explanation for the abnormality is found. The clinical laboratory will clearly mark all laboratory test values that are outside the normal range, and the Investigator will indicate which of these deviations are clinically significant. Clinically significant laboratory result deviations after study drug administration will be recorded as AEs, and the relationship to the treatment will be indicated (see also

Appendix 9.2). Clinically significant laboratory results at screening will not be reported as AE as this is considered part of medical history.

#### 4.5.1.1.9 Vital Signs

Systolic and diastolic blood pressure and pulse will be recorded after the subject has been resting for at least 5 minutes in the supine position. These assessments will be made using an automated device.

## 4.5.1.1.10 Electrocardiogram

A standard 12-lead ECG will be recorded after the subject has been resting for at least 5 minutes in the supine position. The ECG will be recorded using an ECG machine equipped with computer-based interval measurements. The following ECG parameters will be recorded: heart rate, PR-interval, QRS-duration, QT-interval, QTc-interval (Fridericia's), and the interpretation of the ECG profile by the Investigator.

## 4.5.1.1.11 Physical Examination

Physical examination will be performed according to SOPs. In addition, body weight and height will be measured according to SOPs.

### 4.5.1.2 Total of Blood Volume

Table 7 presents the number and volume of blood samples and the total volume of blood that will be collected throughout the study per subject.

If deemed necessary by the Investigator or the Sponsor, the number and/or volume of blood samples per assessment may be increased as long as the total volume of blood drawn for a subject does not surpass 500 mL.

Table 7 Number and Volume of Blood Samples and Total Blood Volume Collected per Subject

| Assessment | Maximum #<br>Samples | Volume of Blood per<br>Sample (mL) | Total Volume of Blood (mL) |
|---|---|---|---|
| Clinical Chemistry | 2 | 3.5 | 7 |
| Hematology | 2 | 3 | 6 |
| Serology | 1 | 5 | 5 |
| Total Volume of Blood Drawn | | | 18 |

### 4.5.2 Appropriateness of Measurements

The assessments that will be made in this study are standard and generally recognized as reliable, accurate, and relevant.

## 4.5.3 Safety Variables

The safety variables to be measured include but are not limited to the variables as given below. A complete list of safety variables will be provided in the statistical analysis plan (SAP).

- Intensity of injection site pain VAS
- Categorical assessment of injection site pain intensity (6-point scale)
- Quality of pain modified SF-MPQ-2 inventory

- Duration of pain
- Comparative pain assessment (5-point scale)
- AEs
- Clinical laboratory (if postdose assessments are deemed relevant by the Investigator)
- Vital signs
- ECG (if postdose assessments are deemed relevant by the Investigator)
- Physical examination (if postdose assessments are deemed relevant by the Investigator)

## 4.6 Statistical Procedures and Determination of Sample Size

## 4.6.1 Analysis Sets

## **4.6.1.1** Safety Set

All subjects who have received at least 1 injection of semaglutide (includes any skin contact with study product whether the injection was completed or not).

## 4.6.1.2 Full analysis set (FAS)

All randomized subjects who have received at least 1 injection of semaglutide (includes any skin contact with trial product whether the injection was completed or not). In exceptional cases, subjects from the FAS may be excluded. In such cases the exclusion will be justified and documented.

#### 4.6.1.3 Per-Protocol Set

All subjects who have received both injections of semaglutide and have completed both intensity of injection site pain assessments.

## 4.6.2 Statistical and Analytical Plan for Safety Evaluation

An SAP will be generated by the Biostatistics Department of the SAP will be finalized prior to database lock. Full details of the analysis to be performed will be included in the SAP.

Any deviation from the SAP will be reported in the section "Changes in Planned Analysis" in the clinical study report (CSR).

## 4.6.2.1 Evaluation of Safety and Tolerability

Safety and tolerability will be assessed through intensity of injection site pain VAS, quality of pain modified SF-MPQ-2 inventory, duration of pain assessment, comparative pain assessment, AEs, clinical laboratory, vital signs, ECGs, and physical examination findings (if results are available after dosing), and any other parameter that is relevant for safety assessment.

## 4.6.2.1.1 Intensity of Injection Site Pain Visual Analogue Scale

The primary endpoint is given in Table 8.

**Table 8** Primary Endpoint

| Endpoint Title | Time Frame | Unit |
|---|---|---|
| Intensity of injection site | 1 min after each injection | mm on a 100 mm horizontal |
| pain | (Day 1) | visual analogue scale |
| | | (where 0 mm = no pain, |
| | | 100 mm = unbearable pain) |

The primary endpoint will be analyzed by a fixed analysis of variance model with VAS score as the dependent variable, and product, injection side (right side, left side), injection number (first injection, second injection), and subject as fixed effects.. From the model, the difference in VAS score between the 2 products is estimated and presented with a 95% CI and a p-value. The interpretation of the difference in VAS pain scores will be supported and contextualized by the results of the analyses of the exploratory endpoints.

# 4.6.2.1.2 Categorical Assessment of Injection Site Pain Intensity, Quality of Pain Modified SF-MPQ-2 Inventory, Duration of Pain, and Comparative Pain Assessment

The exploratory endpoints are given in Table 9.

**Table 9** Exploratory Endpoints

| Endpoint Title | Time Frame | Unit |
|---|---|---|
| Categorical assessment of | Immediately after rating of | 6-point scale (none – very mild |
| injection site pain intensity | intensity of injection site pain, | - mild - moderate - severe - |
| | ie, after 1 min plus the time it | very severe) |
| | takes to complete the rating of | |
| | intensity of injection site pain by | |
| | visual analogue scale (Day 1) | |
| Moderate or more injection site | Dichotomous variable based | Yes = moderate, severe, very |
| pain | on categorical assessment of | severe |
| | intensity of injection site pain | No = none, very mild, mild |
| | (Day 1) (item above) | D : 10 11 |
| Quality of pain | Immediately after categorical | Pain quality items on modified |
| | assessment of intensity of injection site pain, ie, after 1 | SF-MPQ-2 inventory (select all that apply): |
| | min plus the time it takes to | '' '' |
| | complete the rating of intensity | Throbbing pain □ |
| | of injection site pain and the | Shooting pain □ |
| | categorical rating of intensity of | Stabbing pain □ |
| | injection site pain (Day 1) | Sharp pain □ |
| | | Cramping pain □ |
| | | Gnawing pain □ |
| | | Hot-burning pain □ |
| | | Aching pain □ |
| | | Heavy pain □ |
| | | Tender □ |
| | | Splitting pain □ |
| | | Tiring-exhausting □ |
| | | Sickening □ |
| | | Fearful □ |
| | | Punishing-cruel □ |

| Endpoint Title | Time Frame | Unit |
|---|---|---|
| | | Electric-shock pain □ |
| | | Cold-freezing pain □ |
| | | Piercing □ |
| Duration of pain | From time of injection until cessation of pain (Day 1) | min and sec |
| Comparative pain experience | After pain has ended after the last injection (Day 1) | 5-point scale (the last injection hurt much more than the first injection – the last injection hurt more than the first injection – they hurt about the same [includes: none of the injections hurt] – the last injection hurt less than the first injection – the last injection hurt much less than the first injection) |
| The DV3396 product hurt less than or about the same as the PDS290 product | Dichotomous variable based<br>on "Comparative pain<br>experience" variable above<br>(Day 1) | Yes = "about the same (includes none of the products hurt" or "the DV3396 product hurt less than the PDS290 product" or "the DV3396 product hurt much less than the PDS290 product") No= "The DV3396 product hurt much more than the PDS290 product" or "The DV3396 product hurt much more than the PDS290 product hurt more than the PDS290 product" |

The results will be listed, and they will be presented descriptively, where applicable.

#### 4.6.2.1.3 Adverse Events

A listing of all individual AEs will be provided. Summary tables of treatment-emergent adverse events (TEAEs) will be presented by system organ class based on the Medical Dictionary for Regulatory Activities terminology list (preferred terms): one containing the number of TEAEs (frequency of occurrence, number of subjects experiencing the event) by treatment and one containing the number of drug-related TEAEs (frequency of occurrence, number of subjects experiencing the event) per treatment. Additional tables of total counts by treatment and relationship and by treatment and severity will be given.

### 4.6.2.1.4 Technical Complaints

A listing of all technical complaints will be provided.

#### 4.6.2.1.5 Clinical Laboratory

Clinical laboratory data will be listed accompanied by an indication if the parameter is outside the reference range. A summary of all data outside the reference range of the clinical laboratory will be provided. Clinical laboratory data will be presented descriptively, where applicable.

## 4.6.2.1.6 Vital Signs and Electrocardiograms

Vital signs and ECG parameters will be listed, and they will be presented descriptively, where applicable.

#### 4.6.2.1.7 Physical Examination

Changes from baseline for physical examination (if available after dosing) will be described and listed.

## 4.6.3 Determination of Sample Size

The sample size calculation considers both the primary endpoint and the dichotomous endpoints. Considering precision on the proportion of the dichotomous endpoints, a sample size of 100 subjects results in a confidence interval (CI) with a width of 10% on each side, eg, for a proportion of 60%, the CI is 60% (50%-70%).

A standard deviation of within-pair differences in VAS pain score between 2 subcutaneous injections was obtained from Novo Nordisk clinical trial INS-4011. The within-subject variance (adjusting for the effects of speed, volume and injection region) was estimated to 348, corresponding to a standard deviation (SD) of the within-pair difference of  $\sqrt{(2.348)} = 26$  mm. A prospective study of acute pain found that the minimum clinically important difference (MCID) for worsening of pain, ie, the difference on a VAS associated with the selection of "a little more pain" rather than "about the same" had a mean value of 10 mm.<sup>3</sup>

With 100 subjects, a conservative standard deviation of 30 mm, and 90% power, it is possible to detect a difference smaller than 10 mm (Table 10). Hence a sample size of 100 subjects is considered sufficient to detect a clinically important difference. Allowing for 4% dropouts or missing data, a total of 104 subjects will need to be randomized.

Table 10 Detectable Difference with a Sample Size of 100 Subjects for Different Combinations of Power, and Standard Deviation

| Combinations of Fourth and Standard Bottation | | | |
|---|---|---|---|
| Number of | Power | Standard | Difference |
| Subjects | | Deviation | |
| 100 | 0.8 | 25 mm | 7.1 mm |
| 100 | 0.8 | 30 mm | 8.5 mm |
| 100 | 0.9 | 25 mm | 8.2 mm |
| 100 | 0.9 | 30 mm | 9.8 mm |

## 4.6.4 Interim Analysis

After the last subject has completed Day 1, all data collected will be released unblinded for analysis notwithstanding that the subjects have not completed the safety follow-up phone call.

### 4.7 Data Quality Assurance

The study may be audited by the Quality Assurance Department at to assess adherence to the clinical study protocol (CSP) and Quality System. During the conduct of the study, process-related audits may be performed. An audit certificate will be

provided in the appendices of the final CSR outlining any audits and other related activities performed.

The clinical research site will be monitored by the study blinded monitor and unblinded monitor to ensure correct performance of the study procedures and assure that the study is conducted according to the relevant regulatory requirements. The eCRF entries will be verified with the source documentation, if applicable (in some cases there are no source pages, therefore verification is not necessary).

Regulatory authorities, the IEC, and/or the Sponsor's clinical quality assurance group may request access to all source documents, eCRFs, and other study documentation for on-site audit or inspection. Direct access to these documents must be guaranteed by the Investigator, who must provide support at all times for these activities.

Quality control principles will be applied throughout the performance of this study. Review procedures will be followed at for all documents that are generated in relation to the study.

An explanation will be given for all missing, unused, and spurious data in the relevant sections of the CSR.

## 5. ETHICS

## 5.1 Independent Ethics Committee

The CSP and the ICFs will be submitted for review and approval by the IEC of the foundation "Beoordeling Ethiek Biomedisch Onderzoek" (English translation: "Evaluation of Ethics in Biomedical Research") 

The Netherlands) prior to the eligibility screening. The composition of the IEC is in accordance with the recommendations of the World Health Organization, the International Council for Harmonisation (ICH) E6 Guideline for Good Clinical Practice (GCP)<sup>4</sup>, and the EU Clinical Trial Directive (CTD) (Directive 2001/20/EC)<sup>5</sup> (see below).

will keep the IEC informed about the progress of the study. All changes in research activities and all unanticipated problems involving risks to human subjects will be immediately reported to the IEC. In accordance with Section 10, Subsection 1, of the Dutch law on Medical Research in Human Subjects (WMO, revised December 2015)<sup>6</sup>, will inform the subjects and the IEC if anything occurs on the basis of which it appears that the disadvantages of participation may be significantly greater than was foreseen in the research proposal, or if further recruitment of subjects in the study has been put on hold for that reason, whichever occurs first. The study may be suspended pending further review by the IEC, except insofar as suspension would jeopardize the subjects' health.

No changes will be made in the study without IEC approval, except when required to eliminate apparent immediate hazards to human subjects.

Notification of the end of the study will be sent by to the Competent Authority (CA) in The Netherlands and to the IEC within 90 days after completion of follow-up for the last subject. In case a study is temporarily halted, will notify the IEC immediately, including the reason for this. In case a study is ended prematurely, will notify the IEC and the CA in The Netherlands within 15 days, including the reasons for the premature termination. A summary of the results of the study will be sent by to the CA and the IEC within 1 year after the end of the study.

### 5.2 Ethical Conduct of the Study

This study will be conducted in accordance with the ethical principles that have their origin in the World Medical Association (WMA) Declaration of Helsinki, adopted by the 18<sup>th</sup> WMA General Assembly, Helsinki, Finland, June 1964, and subsequent amendments.<sup>7</sup>

This study is also designed to comply with ICH E6 Guideline for GCP (EMA/Committee for Medicinal Products for Human Use [CHMP]/ICH/135/1995)<sup>4</sup> and the EU CTD Directive 2001/20/EC<sup>5</sup>, as incorporated into Dutch Law.<sup>6</sup>

Guidelines adopted by the ICH and other relevant international guidelines, recommendations, and requirements will be taken into account as comprehensively as possible, as long as they do not violate local law.

Whenever the term "Investigator" is noted in the CSP text, it may refer to either the Investigator at the site or an appropriately qualified, trained, and delegated individual of the investigational site.

## 5.3 Subject Information and Consent

All subjects will be informed verbally and in writing regarding the objectives, procedures, and risks of study participation. The subjects will have to sign the Dutch or English version of the ICF before any study-related procedures are started. The ICF contains information about the objectives of the study, the procedures followed during the study, and the risks and restrictions of the study, with special reference to possible side effects of the medication and potential interactions. In addition, insurance coverage provided during the study is explained. The elements addressed in the ICF are according to the ICH E6 Guideline for GCP (EMA/CHMP/ICH/135/1995).<sup>4</sup>

## 5.4 Privacy

All personal details will be treated as confidential by the Investigator and staff at and the handling of personal data will be in compliance with the EU General Data Protection Regulation (GDPR).8

## 6. STUDY ADMINISTRATIVE STRUCTURE

#### 6.1 Distribution of Activities

## Supply of Study Drug

Novo Nordisk A/S Denmark will supply the DV3396 products and the PDS290 products for use in the study.

The PDS290 product will be used with an Ypsomed Clickfine AutoProtect, 8 mm x 29G needle. This needle will be sourced directly by

#### **Laboratory Assessments**

The analysis of clinical laboratory samples will be performed at the Clinical Laboratory.

## eCRF Design

The eCRF design will be performed with the computer program Oracle Clinical by the Database Programming Department of

#### **Data Management**

Data management will be performed with the computer programs Oracle Clinical

by the Data Management Department of ...

#### **Statistics**

An SAP will be generated by the Biostatistics Department of The safety analysis will be conducted by the Biostatistics Department of Statistical analysis will be performed with the computer program SAS (

## **CSR** Writing

The CSR, structured in accordance with the guideline "Structure and Content of Clinical Study Reports - ICH E3", will be written by

## 6.2 Documentation

## 6.2.1 Archiving

All documents concerning the study will be kept on file in the Central Archives of for at least 15 years after conduct of the study. The Sponsor will receive the completed eCRFs (upon request, as PDF file).

## 6.2.2 Recording of Data in Source Documents and eCRFs

Wherever possible, all data will be entered directly into the eCRFs. Source documents will be used in some cases.

A data management plan will be written by the Data Management Department of which will be finalized prior to performing any data validation. An appendix to the data management plan (Origin of Source Data List for Data Entry) will identify any data to be recorded directly in the eCRF (ie, no prior written or electronic record of data) and which data should be considered source data.

## 7. CONFIDENTIALITY AND PUBLICATION POLICY

By signing this CSP, the Investigator reaffirms to the Sponsor that he will maintain in confidence all information furnished to him or resulting from this study. The Investigator will only divulge such information as may be necessary to the IEC, the members of the staff, and the subjects who are involved in this study.

The primary completion date (PCD) is the last assessment of the primary endpoint, and is for this study Day 1. If the last subject is withdrawn early, the PCD is considered the date when the last subject would have completed Day 1. The PCD determines the deadline for results disclosure at clinicaltrials.gov according to the Food and Drug Administration Amendments Act.

## 7.1 Publication Policy

Novo Nordisk commits to communicate and disclose results of trials regardless of outcome. Disclosure includes publication of a manuscript in a peer-reviewed scientific journal, abstract submission with a poster or oral presentation at a scientific meeting or disclosure by other means. The results of this trial will be subject to public disclosure on external web sites according to international and national regulations. Novo Nordisk reserves the right to defer the release of data until specified milestones are reached, for example when the clinical trial report is available. This includes the right not to release the results of interim analyses, because the release of such information may influence the results of the entire trial. At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 30 days to protect intellectual property. In all cases the trial results will be reported in an objective, accurate, balanced and complete manner, with a discussion of the strengths and limitations. In the event of any disagreement on the content of any publication, both the investigators' and Novo Nordisk opinions will be fairly and sufficiently represented in the publication.

#### 7.2 Dissemination of Clinical Trial Data

Information of the trial will be disclosed at clinicaltrials.gov and novonordisk-trials.com. It will also be disclosed according to other applicable requirements such as those of the International Committee of Medical Journal Editors, the Food and Drug Administration Amendments Act, European Commission Requirements, and other relevant recommendations or regulations. If a subject requests to be included in the trial via the Novo Nordisk e-mail contact at these websites, Novo Nordisk may disclose the Investigator's contact details to the subject. As a result of increasing requirements for transparency, some countries require public disclosure of Investigator names and their affiliations.

## 8. REFERENCES

- 1. Novo Nordisk A/S. Investigator's Brochure, semaglutide s.c. for weight management and non-alcoholic steatohepatitis, projects NN9536 and NN9931 (edition 4). Mar 2019.
- Dworkin RH, Turk DC, Revicki DA, et al. Development and initial validation of an expanded and revised version of the Short-form McGill Pain Questionnaire (SF-MPQ-2). Pain. 2009;144:35-42.
- 3. Todd KH, Funk KG, Funk JP, et al. Clinical significance of reported changes in pain severity. Ann Emerg Med.1996;27:485-89.
- International Council for Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonised Tripartite Guideline, E6 (R2): Guideline for Good Clinical Practice (EMA/CHMP/ICH/135/1995), 15 December 2016.
- 5. Directive 2001/20/EC of the European Parliament and of the Council of 4 April 2001 on the approximation of the laws, regulations and administrative provisions of the Member States relating to the implementation of good clinical practice in the conduct of clinical trials on medicinal products for human use.
- 6. Medical Research Involving Human Subjects Act (WMO, Wet Medisch-Wetenschappelijk Onderzoek met Mensen), revision December 2015.
- 7. WMA Declaration of Helsinki (18th WMA General Assembly 1964), revised at 64th World Medical Association General Assembly, Fortaleza, Brazil, October 2013.
- 8. The General Data Protection Regulation (GDPR). Regulation (EU) 2016/679 of the European Parliament and the Council of the European Union, 27 April 2016.
- 9. International Council for Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonised Tripartite Guideline, E3: Structure and Content of Clinical Study Reports (CPMP/ICH/137/95), November 1995.
- International Council for Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonised Tripartite Guideline, E2A: Clinical Safety Data Management: Definitions and Standards for Expedited Reporting, Note for Guidance on Clinical Safety Data Management, June 1995.

## 9. APPENDICES

## 9.1 Drug Accountability

- Study product storage, in-use conditions and in-use time will be available on the label and in the TMM. The Investigator must confirm that appropriate temperature conditions have been maintained during transit for all study products received and any discrepancies are reported and resolved before use of the study products.
- All study products must be stored in a secure, controlled, and monitored (manual or automated) area in accordance with the labelled storage conditions with access limited to the pharmacist and pharmacy assistant.
- The Investigator must inform Novo Nordisk immediately if any study product has been stored outside specified conditions. Additional details regarding handling of temperature deviations can be found in the TMM.
- Study product that has been stored improperly must not be dispensed to any subject before it has been evaluated and approved for further use by Novo Nordisk.
- The Investigator is responsible for drug accountability and record maintenance (ie, receipt, accountability and final disposition records).
- For study products packed unblinded in a blinded study: Drug accountability will be performed by an unblinded person who will ensure that unblinding information such as batch numbers are not revealed to personnel that should remain blinded).
- Drug accountability should be performed at dose level unless this is not possible (eg, products in pen-injectors), then describe and explain the actual level of accountability.

# 9.2 Adverse Events: Definitions and Procedures for Recording, Evaluation, Follow-up, and Reporting to Sponsor

#### AE definition

- An AE is any untoward occurrence in a clinical trial subject that is temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
- An AE can be any unfavorable and unintended sign, including an abnormal laboratory finding, symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.

#### **Events meeting the AE definition**

- Any abnormal laboratory test results or safety assessments, including those that worsen
  from baseline, considered clinically significant in the medical and scientific judgment of the
  investigator.
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of trial product regardless of intent.

## **Events NOT** meeting the AE definition

 Pre-existing conditions, anticipated day-to-day fluctuations of pre-existing conditions, including those identified during screening or other trial procedures performed before exposure to trial product.

Note: Pre-existing conditions should be recorded as medical history/concomitant illness.

- Pre-planned procedures, unless the condition for which the procedure was planned has worsened from the first trial-related activity after the subject has signed the informed consent.
- Pain: Non-serious pain will be collected on specific pain-rating schemes please refer to
  the schedule of assessments (Table 1) and Section 4.5.
   If the event of pain fulfils the criteria for an SAE then in addition to the above, an AE form
  and a safety information form must also be filled in.

#### Definition of an SAE

#### An SAE is an AE that fulfils at least one of the following criteria:

#### · Results in death

#### Is life-threatening

The term 'life-threatening' in the definition of 'serious' refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event which hypothetically might have caused death, if it were more severe.

## • Requires inpatient hospitalisation or prolongation of existing hospitalisation

- Hospitalization signifies that the subject has been detained at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalisation are AEs. If a complication prolongs hospitalization or fulfils any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.
- Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

#### Note:

- Hospitalizations for administrative, trial-related and social purposes do not constitute AEs and should therefore not be reported as AEs or SAEs.
- Hospital admissions for surgical procedures, planned before trial inclusion, are not considered AEs or SAEs.

## · Results in persistent disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experience of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhoea, influenza, and accidental trauma (eg, sprained ankle), which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### Is a congenital anomaly/birth defect

· Including events leading to fetal distress or fetal death

#### • Important medical event:

- Medical or scientific judgment should be exercised in deciding whether SAE reporting
  is appropriate in other situations. This includes important medical events that may not
  be immediately life-threatening or result in death or hospitalization, but may jeopardize
  the subject or may require medical or surgical intervention to prevent one of the other
  outcomes listed in the above definition. These events should usually be considered
  serious and reported as SAEs using the important medical event criterion.
- The following AEs must always be reported as SAEs using the important medical event criterion, if no other seriousness criteria are applicable:
  - suspicion of transmission of infectious agents via the trial product.
  - risk of liver injury defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 x the upper limit of normal (ULN) and total bilirubin >2 x ULN, where no alternative etiology exists (Hy's law).
  - events that might have led to or might lead directly or indirectly to death or a serious deterioration in state of health

These are handled under the SAE reporting system.

## Description of AEs requiring additional data collection (via specific event form)

#### Medication error:

A medication error concerning trial products is defined as:

- Administration of wrong drug or use of wrong device.
   Note: Use of wrong DUN is not considered a medication error unless it results in a confirmed administration of wrong drug.
- Wrong route of administration, such as intramuscular instead of sc
- Accidental administration of a lower or higher dose than intended. The administered dose
  must deviate from the intended dose to an extent where clinical consequences for the trial
  subject were likely to happen as judged by the investigator, although they did not
  necessarily occur.

#### AE and SAE recording

- The investigator will record all relevant AE information in the eCRF and SAE information on paper forms.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. In such cases, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.
- When an AE/SAE occurs, it is the responsibility of the investigator to review all documentation (eg, hospital progress notes, laboratory and diagnostics reports) related to the event.
- For all non-serious AEs the applicable forms should be signed when the event is resolved
  or at the end of the trial at the latest. For sign-off of SAE-related forms, refer to "SAE
  reporting via paper CRF" later in this section.
- Novo Nordisk products used as concomitant medication: if an AE is considered to have a
  causal relationship with a Novo Nordisk marketed product used as concomitant
  medication in the trial, it is important that the suspected relationship is reported to Novo
  Nordisk, eg, in the alternative etiology section on the safety information form. Novo
  Nordisk may need to report this adverse event to relevant regulatory authorities.

#### Assessment of severity

The investigator will assess intensity for each event reported during the trial and assign it to one of the following categories:

- **Mild**: An event that is easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities.
- Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities.
- Severe: An event that prevents normal everyday activities.
   Note: Severe is a category used for rating the intensity of an event; and both an AE and SAE can be assessed as severe. An event is defined as 'serious' when it meets at least one of the outcomes described in the definition of an SAE and not when it is rated as severe.

#### Assessment of causality

The investigator is obligated to assess the relationship between trial product and the occurrence of each AE/SAE.

Relationship between an AE/SAE and the relevant trial product(s) should be assessed as:

- Probable Good reason and sufficient documentation to assume a causal relationship.
- Possible A causal relationship is conceivable and cannot be dismissed.
- Unlikely The event is most likely related to etiology other than the trial product. Alternative etiology, such as underlying disease(s), concomitant medication, and other risk factors, as well as the temporal relationship of the event to trial product administration will be considered and investigated.

The investigator should use the investigator's brochure for the assessment. For each AE/SAE, the investigator must document in the medical records that he/she has reviewed the AE/SAE and has provided an assessment of causality.

There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report. However, it is important that the investigator always makes an assessment of causality for every event before the initial transmission of the SAE data.

The investigator may change his/her opinion of causality in light of follow-up information and send a follow-up report with the updated causality assessment.

The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### Final outcome

The investigator will select the most appropriate outcome:

- **Recovered/resolved**: The subject has fully recovered, or by medical or surgical treatment the condition has returned to the level observed at the first trial-related activity after the subject signed the informed consent.
- Recovering/resolving: The condition is improving, and the subject is expected to recover from the event. This term is only applicable if the subject has completed the trial or has died from another AE.
- Recovered/resolved with sequelae: The subject has recovered from the condition, but
  with lasting effect due to a disease, injury, treatment, or procedure. If a sequelae meets
  an SAE criterion, the AE must be reported as an SAE.
- **Not recovered/not resolved**: The condition of the subject has not improved and the symptoms are unchanged or the outcome is not known.
- Fatal: This term is only applicable if the subject died from a condition related to the
  reported AE. Outcomes of other reported AEs in a subject before he/she died should be
  assessed as "recovered/resolved," "recovering/resolving," "recovered/resolved with
  sequelae," or "not recovered/not resolved." An AE with a fatal outcome must be reported
  as an SAE.
- Unknown: This term is only applicable if the subject is lost to follow-up.

## Follow-up of AE and SAE

The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by Novo Nordisk to elucidate the nature and/or causality of the AE or SAE as fully as possible (eg, severe hypersensitivity reactions). This may include additional laboratory tests (eg, skin prick test) or investigations, histopathological examinations, or consultation with other health care professionals.

If a subject dies during participation in the trial or during a recognized follow-up period, the investigator should provide Novo Nordisk with a copy of autopsy report including histopathology.

New or updated information will be recorded in the CRF.

#### SAE reporting via paper CRF

- Relevant CRF forms (AE and safety information forms) must be forwarded to Novo Nordisk.
- The Investigator needs to complete the AE and safety information form within the designated reporting time frames (as illustrated in Figure 2).
- If the eCRF is unavailable for more than 24 hours, then the site will use the paper AE form.

Contact details for SAE reporting can be found in the investigator trial master file.

## **Memo to File**

| То: | File |
|-------|------------------|
| From: | |
| Date: | |
| RE: | Site Affiliation |

## The following Investigators are affiliated with



| Name | Signature | Date (dd-Mmm-yyyy) |
|------|-----------|--------------------|